CLINICAL TRIAL: NCT02255669
Title: Comparison Between Fully Covered and Partially Covered Self-expandable Metal Stents With Anti-migration System for Malignant Distal Biliary Obstruction
Brief Title: Fully Covered SEMS Versus Partially Covered SEMS With Anti-migration System for Malignant Distal Biliary Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-07-187-001
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2014-09

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- partially covered SEMS (Active Comparator): Deployment of Partially covered biliary self expandable metal stent
  Interventions: Device: partially covered SEMS
- fully covered SEMS (Active Comparator): Deployment of Fully covered biliary self expandable metal stent
  Interventions: Device: fully covered SEMS

INTERVENTIONS:
Device: partially covered SEMS — Used for palliation of inoperable malignant distal bile duct obstruction.
  Other Names: Insertion of partially covered SEMS (PCSEMS)
  Arms: partially covered SEMS
Device: fully covered SEMS — Used for palliation of inoperable malignant distal bile duct obstruction.
  Other Names: Insertion of fully covered SEMS (FCSEMS)
  Arms: fully covered SEMS

SUMMARY:
The purpose of this study is to compare the duration of stent patency between partially covered and fully covered SEMS for palliation of malignant distal bile duct obstruction.

DETAILED DESCRIPTION:
Endoscopic stent placement has been used as a principle palliative method in patients with unresectable distal malignancy biliary obstruction. It has been pivotal in providing relief from obstructive jaundice, improving the quality of life, and allowing the maintenance of chemotherapy. Although SEMSs have been reported to be superior to plastic stents in terms of stent patency, they still have some debatable issues ; in uncovered SEMS, stent occlusion due to epithelial hyperplasia and tumor ingrowth through the metal mesh is a frequent problem, whereas covered SEMSs are prone to migration.

The aim of the current study is to compare the duration of stent patency between partially covered and fully covered SEMS as a primary objective, and investigate overall patient survival, stent occlusion rate, and incidence of adverse events including stent dysfunction as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* 1.> 19years 2.malignant biliary obstruction, 2 cm distal to hilum 3.unsuitable for curative surgical resection owing to metastasis, locally advanced stage, high operation risk, or patient's refusal

Exclusion Criteria:

* 1.history of biliary surgery except cholecystectomy 2.history of SEMS placement 3.coagulopathy (INR>1.5, Platelet<50000) 4.expected survival > 3 months based on Karnofsky performance score 5.duodenal stricture

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
duration of stent patency | From the date of randomization until the date of first documented stent dysfunction, assessed upto 12 months

SECONDARY OUTCOMES:
overall survival | From the date of randomization until the date of death from any cause, assessed upto 12 months
stent occlusion rate | From the date of randomization until the date of first documented stent occlusion, assessed up to 12 months
stent related complication | From the date of randomization until the date of first documented stent related complication, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jong Kyun Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Cencer
Locations (1):
- Samsung Medical Cencer, Seoul, South Korea